CLINICAL TRIAL: NCT03589053
Title: Effects of Limb Remote Ischemic Conditioning (LRIC) on Cerebrovascular Reserve (CVR) in Ischemic Cerebrovascular Disease Patients
Brief Title: Limb Remote Ischemic Conditioning and Cerebrovascular Reserve
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRIC-CVR
Record Dates: First submitted 2018-06-28; First posted 2018-07-17 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Ischemic Cerebrovascular Disease
Keywords: Limb remote ischemic conditioning; Cerebrovascular reserve
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LRIC group (Experimental): Participants in the experimental group receive both LRIC and standard clinical therapy. The LRIC treatment is composed of 5 cycles of bilateral upper limb ischemia for 5 minutes followed by reperfusion for another 5 minutes performed twice a day for a total of 90 consecutive days.The procedure was performed by using an electric autocontrol device with cuffs that inflated to a pressure of 200 mmHg during the ischemic period and deflated during the reperfusion (Patent No.CN200820123637.X, China).
  Interventions: Device: Limb remote ischemic conditioning
- Control group (Sham Comparator): Participants in the control group receive both sham LRIC and standard clinical therapy.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Limb remote ischemic conditioning — The LRIC treatment consisted of 5 cycles of bilateral upper limb ischemia for 5 minutes followed by reperfusion for another 5 minutes performed twice a day for a total of 90 consecutive days.The procedure was performed by using an electric autocontrol device with cuffs that inflated to a pressure of 200 mmHg during the ischemic period and deflated during the reperfusion.
  Arms: LRIC group
Device: Control group — Participants in the control group receive both sham LRIC and standard clinical therapy.
  Arms: Control group

SUMMARY:
Cerebrovascular reserve (CVR), defined as the increase in cerebral blood flow (CBF)in response to a vasodilatory stimulus, is known to reflect the compensative capacity of the brain to maintain adequate blood flow in the face of decreased perfusion due to arterial stenosis. CVR dysfunction has been identified as an independent risk factor for ischemic stroke. Limb remote ischemic preconditioning （LRIC) has been suggested as a protective therapeutic modality against brain ischemia. So it is worth to detect whether LRIC can improve the CVR ability in ischemic cerebrovascular disease patients.

ELIGIBILITY:
Inclusion Criteria:

- (1)Symptomatic intracranial arterial stenosis measuring >=50% by angiography or >=70% by ultrasound, CT angiography (CTA), or magnetic resonance angiography (MRA);(2)Age range 18-80 years;(3)Compared with normal brain tissue, the reduction of cerebral glucose metabolism (CGM) and/ or cerebral blood flow (CBF) in the focal area>=8%;(4)Stable vital signs, normal renal and hepatic functions; (5)No hemorrhagic tendency;(6)Subject or his or her legally authorized representative was able to provide an informed conised.

Exclusion Criteria:

-(1)Uncontrolled hypertension (defined as systolic blood pressure>=200 mmHg despite medications at enrollment); (2)Any vascular, soft tissue, or orthopedic injury (eg, superficial wounds and fractures of the arm) that contraindicated bilateral arm ischemic preconditioning;(3)Peripheral vascular disease (especially subclavian arterial and upper limb artery stenosis or occlusion); (4)Hematologic disease;(5)Severe or unstable concomitant disease;(6)Can not tolerate LRIC treatment;(7)No informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-08 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of cerebrovascular reserve | 90 days
  We evaluate the compensatory capacity of cerebral blood vessels and brain tissue by the rate of changes in cerebral blood flow and brain metabolism under stress and resting conditions, respectively.

SECONDARY OUTCOMES:
Recurrence of stroke | 90 days

OTHER OUTCOMES:
Safety of LRIC [Number of patients not tolerating RIC procedure and patients with erythema or skin lesions related to RIC] | 90 days
  The safety of LRIC by the number of patients not tolerating RIC procedure and patients with erythema or skin lesions related to RIC.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Principal Investigator — Capital Medical University
Locations (1):
- Xunming Ji, Beijing, Beijing Municipality, China